CLINICAL TRIAL: NCT04591314
Title: Evaluation of the Effect of Neurofeedback Targeting EEG Theta / Beta Activities on the Strengthening of Wakefulness Maintenance Capacities and Cognitive Performance.
Acronym: NEUROWAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2020/28
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Sleep Deprivation
Keywords: Neurofeedback; electroencephalography; sleep deprivation; maintenance wakefulness test; cognitive performance; learning modulation; arousal system.
MeSH Terms: conditions — Sleep Deprivation | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback participants (Experimental): All the participants studied.
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — The intervention by neurofeedback (NF) will consist in providing the subjects with a feedback on their EEG Theta / Beta activity in real time Each subject will perform 8 sessions of neurofeedback (1h30 / session, 40 min of effective training by neurofeedback) at an average rate of 1 to 2 sessions per week.

SUMMARY:
Neurofeedback is a cognitive remediation technique that allows a subject to learn to regulate their cognitive and brain activity through information provided in real time about their brain activity, in particular electroencephalographic (EEG) brain activity. Neurofeedback could, through its impact on the degree of neuronal synchronization, help to reduce the impact of sleep deprivation on wakefulness and cognitive performance. The main objective is to study the effect of a program of 8 sessions of neurofeedback targeting EEG theta / beta activities, to modify the degree of neuronal synchronization, on the ability to maintain objective wakefulness measured by a maintenance wakefulness test (MWT) in healthy subjects presenting objective excessive daytime sleepiness after a full night of sleep deprivation under controlled experimental conditions. The objective of this study will also provide a better understanding of the learning modulation mechanisms of arousal systems.

DETAILED DESCRIPTION:
Neurofeedback is a cognitive remediation technique that allows a subject to learn to regulate their cognitive and brain activity through information provided in real time about their brain activity, in particular electroencephalographic (EEG) brain activity. Neurofeedback has been used to regulate EEG amplitude in certain spectral bands, which correlate with the degree of neural synchronization. Neurofeedback makes it possible in particular to reduce the amplitude of the EEG theta spectral band (4-8 Hz) and to increase the EEG beta spectral band (> 12Hz).

This type of protocol has been used successfully to reduce the degree of neural synchronization and to stimulate arousal systems and sustained attention skills.

Studies on healthy subjects submitted to controlled sleep deprivation have shown that inducing a full night of sleep deprivation is a good model for studying the brain mechanisms of arousal and the links with cognitive functions, but also to assess the effectiveness of counter measures reducing the impact of sleep deprivation on cognitive performance. These experimental models provide a better understanding of the mechanisms and consequences of the complaint of excessive daytime sleepiness (EDS). EDS is indeed a frequent symptom affecting between 5% and 8% of the population. The consequence of EDS is a decrease in quality of life. In addition, the EDS entails a high medico-economic cost because of the accidental risk of the public and professional roads.

Neurofeedback could, through its impact on the degree of neuronal synchronization, help to reduce the impact of sleep deprivation on wakefulness and cognitive performance. Thus, it appears relevant to assess the effectiveness of neurofeedback, targeting activities in the theta / beta EEG spectral band, on wakefulness and cognitive performance in healthy subjects with EDS due to sleep deprivation. Targeting the degree of neuronal EEG synchronization would then be an innovative avenue for improving the physiological mobilization of arousal systems and wakefulness and cognitive performance in the event of EDS. This cognitive remediation technique could in particular be proposed as a complement to pharmacological treatment in treated patients suffering from hypersomnolence disorder presenting a residual EDS.

The main objective is to study the effect of a program of 8 sessions of neurofeedback targeting EEG theta / beta activities, to modify the degree of neuronal synchronization, on the ability to maintain objective wakefulness measured by a maintenance wakefulness test (MWT) in healthy subjects presenting objective excessive daytime sleepiness after a full night of sleep deprivation under controlled experimental conditions. The objective of this study will also provide a better understanding of the learning modulation mechanisms of arousal systems.

The secondary objectives are:

1. To study the effect of a program of 8 sessions of neurofeedback targeting theta / beta EEG activities, in healthy subjects after a full night of sleep deprivation presenting objective excessive daytime sleepiness, on the instantaneous subjective arousal level in a situation controlled (MWT and neurofeedback session) by the Karolinska sleepiness scale (KSS).
2. To study the effect of a program of 8 sessions of neurofeedback targeting theta / beta EEG activities, in healthy subjects after a full night of sleep deprivation presenting objective excessive daytime sleepiness, on the cognitive performance, before and after neurofeedback sessions, assessed by the Psychomotor Vigilance Task (PVT) and by the Test of Attentional Performance (TAP).
3. To study the functional reorganization of the EEG activities of the brain, in particular the degree of neuronal synchronization between the different regions of the scalp, in subjects presenting objective excessive daytime sleepiness after a full night of sleep deprivation and following a program of 8 neurofeedback sessions targeting EEG theta / beta activities.
4. To study a learning effect during the 8 neurofeedback sessions evaluated by measuring the evolution of the modulation of the spectral power in the theta / beta band during each neurofeedback session.
5. To study the prognostic learning factors during the 8 neurofeedback sessions.
6. To study the prognostic factors for clinical improvement of MWT, subjective EDS and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 35 years old,
* Healthy subject, no pathology reported at the interview
* Absence of EDS complaints (total ESS score<11) and sleep complaints (total Insomnia Severity Indexscore <15)
* Presence of an objective EDS measured by a mean sleep latency of less than 30 minutes on the wakefulness maintenance test performed after a night of total sleep deprivation under controlled conditions (at the inclusion visit),
* Motivated to carry out the program of 8 neurofeedback sessions,
* Body mass index < 25 kg/m2,
* Affiliated with the social security (beneficiary or entitled person),
* Having been informed and having signed an informed consent.

Exclusion Criteria:

* All pathologies that may induce excessive daytime sleepiness: untreated narcolepsy or idiopathic hypersomnia, untreated sleep apnea syndrome, untreated restless legs syndrome, untreated periodic leg movement syndrome, unstabilized psychiatric disorders of the characterized depressive disorder type, anxiety disorders, bipolar disorder, addictive disorders (alcohol and drugs), obesity having undergone surgical treatment for less than 3 months.
* Chronic insomnia disorder
* Excessive consumption of coffee, tea, or caffeinated cola type beverages (> 5 cups/day)
* All pathologies making interaction with the neurofeedback device potentially problematic: intellectual, visual, auditory or motor impairment, psychotic disorders, unstable cardio-respiratory diseases, neurological disease of the central nervous system, confusion, dementia,
* Any situation or treatment modifying the EEG spectral power: psychotropic treatments, night or shift work, chrono-biological disorders interfering with the level of daytime alertness, history of cranial surgery, epilepsy,
* Pregnant or breastfeeding woman,
* Persons placed under the safeguard of justice,
* A person participating in another research study with an exclusion period still in progress,
* Person whose physical and/or psychological health is severely impaired

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Maintenance Wakefulness Test | 1 week after the end of the neurofeedback program (6 weeks after inclusion [day 0])
  Mean latency on the Maintenance Wakefulness Test (MWT) after a full night of sleep deprivation.

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale | At inclusion [day 0], each neurofeedback sessions (weeks 1,2,3,4,5), and 1 week after the end of the neurofeedback program (6 weeks after inclusion [day 0])
  Subjective daytime wakefulness level. minimum value 1 (extremely alert); maximum value 9 (extremely sleepy, fighting sleep)
Cognitive performance (1) | At inclusion [day 0] and 1 week after the end of the neurofeedback program (6 weeks after inclusion [day 0])
  Psychomotor Vigilance Task (PVT),
Cognitive performance (2) | At inclusion [day 0] and 1 week after the end of the neurofeedback program (6 weeks after inclusion [day 0])
  Test of Attention Performance (TAP)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No